CLINICAL TRIAL: NCT06853873
Title: Counseling for Alcohol Problems in Pregnancy (CAP-Pre) Phase II
Acronym: CAP-Pre
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Leibniz Institute for Prevention Research and Epidemiology - BIPS GmbH (Other)
Collaborators: Technical University of Munich (Other); Medical Research Council, South Africa (Other)
Responsible Party: Principal Investigator, Daniela C. Fuhr, Prof, Leibniz Institute for Prevention Research and Epidemiology - BIPS GmbH
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 01KA2401A
Record Dates: First submitted 2025-02-25; First posted 2025-03-03 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Alcohol Use Disorder
Keywords: Alcohol misuse; pregnancy; Women; Psychoeducation; Lay Health Workers; South Africa; Alcohol use in Pregnancy; Counseling Sessions; Psychoeducational Intervention
MeSH Terms: conditions — Alcoholism | interventions — Ethanol; Pregnancy; Methods

STUDY DESIGN:
Intervention Model Description: The study follows a parallel-arm, individually randomized controlled trial (RCT) design to assess the feasibility, acceptability, and preliminary effectiveness of the Counselling for Alcohol Problems in Pregnancy (CAP-Pre) intervention. Participants (n=40 pregnant women, ≤28 weeks gestation) will be randomly assigned (1:1) to either:
  Intervention Group: CAP-Pre plus Enhanced Usual Care (EUC), consisting of five manualized counselling sessions delivered by trained community health workers (CHWs).
  Control Group: EUC only, including an information booklet on alcohol use in pregnancy but no structured counselling.
  Primary outcomes focus on alcohol consumption, measured via self-report (TLFB). Secondary outcomes assess biomarkers for alcohol consumption PeTH testing, psychosocial functioning (WHO-DAS), depressive symptoms (EPDS), alcohol-related consequences (AUDIT-C) and perceived usefulness (qualitative interviews). Data will be collected at baseline and intervention
Who Masked: Investigator, Outcomes Assessor
Masking Description: This study employs single-blind masking, where participants and intervention providers (community health workers) are aware of group assignments. Data collectors and assessors conducting follow-up evaluations are blinded to treatment allocation. This ensures objective data collection and reduces potential observer bias in outcome assessments. To maintain blinding, assessors will not be involved in intervention delivery and will not have access to participant allocation records.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced Usual Care (EUC) (No Intervention): Information booklet on alcohol use in pregnancy. Referral to antenatal services if needed. No structured counseling was provided.
- CAP-Pre + Enhanced Usual Care (Experimental): The Counselling for Alcohol Problems in Pregnancy (CAP-Pre) intervention
  Interventions: Behavioral: The Counselling for Alcohol Problems in Pregnancy (CAP-Pre) intervention

INTERVENTIONS:
Behavioral: The Counselling for Alcohol Problems in Pregnancy (CAP-Pre) intervention — Five structured 60-minute counseling sessions (weekly, CHW-delivered).
  Key components:
  Motivational interviewing (MI) to enhance behavior change. Cognitive-behavioral strategies (CBT) for managing alcohol cravings. Goal-setting and self-monitoring for tracking progress. Problem-solving techniques and social support enhancement.
  Other Names: CAP-PRE
  Arms: CAP-Pre + Enhanced Usual Care

SUMMARY:
Purpose: This study is testing a new counseling program called Counselling for Alcohol Problems in Pregnancy or CAP-Pre, designed to help pregnant women in South Africa to reduce their alcohol use and improve their well-being. Alcohol use during pregnancy can harm babies, leading to Fetal Alcohol Spectrum Disorders (FASD), which can cause lifelong health and developmental problems. Currently, there are no community-based support programs to help pregnant women struggling with alcohol use.

What Happens in the Study? 40 pregnant women will take part in the study and will be randomly assigned to one of two groups:

1. CAP-Pre + Standard Health Advice - Women will receive five counseling sessions to help them reduce drinking, plus usual pregnancy care.
2. Standard Health Advice Only - Women will receive usual pregnancy care and an information booklet on alcohol use in pregnancy.

The study will test:

The study will evaluate if CAP-Pre is easy to deliver, acceptable, and helps women to drink less. (measured by self-report and a blood test).

Why Is This Important? South Africa has the highest rates of FASD in the world, but most pregnant women do not receive specialized support for harmful alcohol use. If this pilot study is successful, it will help prepare for a more extensive study to test whether CAP-Pre can be widely used in antenatal care programs.

Who Is Involved? The study is run by researchers from Germany and South Africa, with funding from the German Alliance for Global Health Research.

DETAILED DESCRIPTION:
South Africa has the highest prevalence of Fetal Alcohol Spectrum Disorders (FASD) globally, with alcohol use during pregnancy being prevalent in low-resource settings. However, there is no structured, community-based psychological support available for pregnant women who consume alcohol at harmful levels. The Counselling for Alcohol Problems in Pregnancy (CAP-Pre) intervention is a brief psychological counseling program designed to:

* Support pregnant women in reducing alcohol use through motivational interviewing (MI) and cognitive-behavioral techniques (CBT).
* Improve maternal well-being by addressing underlying stressors and barriers to change.
* Be delivered by community health workers (CHWs) in a scalable, task-shifted approach.

This pilot randomized controlled trial (RCT) aims to evaluate the CAP-Pre intervention's perceived effectiveness, feasibility, and acceptability in preparation for a definitive RCT.

Study Design Type: Parallel-arm, single-blind, individually randomized controlled trial (RCT).

Setting: Community-based antenatal care program, Cape Flats, Western Cape, South Africa.

Participants: 40 pregnant women screened for the following eligibility criteria

Inclusion:

* ≥18 years old, ≤28 weeks pregnant.
* AUDIT score 8-20 (indicating hazardous alcohol use).

Exclusion:

* Severe psychiatric disorders.
* High-risk pregnancy complications. Recruitment Sites: Community outreach and antenatal clinics.

Randomization: 1:1 allocation to:

* CAP-Pre + Enhanced Usual Care (EUC) (Intervention)
* Enhanced Usual Care (EUC) only (Control) Intervention and Control Groups Intervention: CAP-Pre + Enhanced Usual Care (EUC) (n=20) Five structured 60-minute counseling sessions (weekly, CHW-delivered).

Key components:

Motivational interviewing (MI) to enhance behavior change. Cognitive-behavioral strategies (CBT) for managing alcohol cravings. Goal-setting and self-monitoring for tracking progress. Problem-solving techniques and social support enhancement. Control: Enhanced Usual Care (EUC) (n=20) Information booklet on alcohol use in pregnancy. Referral to antenatal services if needed. No structured counseling was provided.

Data Collection and Outcome Measures

Data Collection Timeline:

Baseline assessment before randomization and Post-intervention assessment on alcohol use, mental health, and qualitative feedback Primary Outcomes

Reduction in alcohol consumption measured through:

Self-Reported Alcohol Use: Alcohol consumption will be assessed using the Alcohol Timeline Follow Back (TLFB) method to estimate daily drinking volume over the past months.

Secondary Outcomes

1. Biological Markers for alcohol consumption: Phosphatidyl ethanol (PeTH) through Dried Blood Spot (DBS) Collection. PeTH is a direct biomarker of alcohol consumption that is formed only in the presence of ethanol. It is highly specific and sensitive in detecting alcohol use over the past 2-3 weeks.
2. Psychosocial Functioning: Assessed using the WHO-Disability Assessment Schedule (WHO-DAS). WHO-DAS 2.0 is a standardized instrument developed by the World Health Organization (WHO) to assess functional impairment and disability across multiple life domains. It evaluates the impact of mental and physical health conditions on daily activities and social participation.
3. Depressive Symptoms: Evaluated using the Edinburgh Postnatal Depression Scale (EPDS). EPDS is a 10-item self-report measure designed to screen for perinatal depression in pregnant and postpartum women.
4. Alcohol-Related Consequences: Measured with the Alcohol Use Disorder Identification Test - Consumption (AUDIT-C). AUDIT-C is a brief, 3-item screening tool derived from the full 10-item Alcohol Use Disorders Identification Test (AUDIT) to identify individuals at risk for hazardous drinking and alcohol use disorders (AUDs).
5. Family and Social Support: Assessed using a 10-item structured questionnaire measuring the availability and perceived adequacy of social support across various domains, such as emotional, instrumental, and informational support.
6. Perceived Usefulness of Counselling: Evaluated through qualitative pre and post-intervention interviews, exploring participant expectations, experiences, perceptions of counseling, and perceived benefits or challenges.

Baseline Covariates:

Additional Covariates Collected at Baseline

1. Demographic and Socioeconomic Information: Age, education, and socioeconomic status.
2. Substance Use and Risk Factors: Self-reported past-month use of tobacco and other substances.
3. Partner Substance Use: Self-reported data on household and partner alcohol/drug use.
4. Intimate Partner Violence (IPV) & History of Trauma: Self-reported experiences of violence, abuse, and health-related risks.
5. Childhood Adversity and Life Stressors: Self-reported early trauma and current stressors.

Analysis Plan We will analyze and report data following CONSORT guidelines for pilot and feasibility trials. Analyses for the pilot RCT will mainly be descriptive to describe recruitment and response rates, process data, and retention at 3 months.

Ethical Considerations This study poses minimal risks, including minor discomfort from blood sampling and potential mental distress during sessions. Confidentiality will be protected through strict data security, staff confidentiality agreements, and ethical training. PeTH blood collection will follow infection control protocols and be conducted by trained staff. Mental distress risks will be minimized through participant choice, referrals for support, and staff supervision. The study has ethical approval from the South African MRC, and participation is voluntary, with the right to withdraw at any time.

Output A contextually adapted program of care (called CAP-PRE) for pregnant women who misuse alcohol that can be tested for effectiveness and cost-effectiveness in a larger, definitive RCT.

ELIGIBILITY:
Inclusion Criteria:

* • Pregnant women ≤28 weeks gestation.

  * Alcohol Use Risk: Hazardous alcohol use, defined as an Alcohol Use Disorder Identification Test (AUDIT) score of 8-20.
  * Age ≥18 years old at the time of recruitment.
  * Consent: Ability to provide written informed consent and willingness to participate in the study

Exclusion Criteria:

* Severe Mental Health Conditions: Diagnosed psychotic disorders or severe cognitive impairment that may interfere with participation.

High-Risk Pregnancy: Presence of significant pregnancy complications that require specialized medical care.

Substance Dependence (Other Than Alcohol): Current dependence on drugs other than alcohol and tobacco requiring specialized treatment.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — This study exclusively includes pregnant women (gender females) who are ≤28 weeks gestation at the time of recruitment. The rationale for this gender-based inclusion is that pregnancy-related alcohol consumption and its associated risks, such as Fetal Alcohol Spectrum Disorders (FASD), are biologically specific to individuals who can become pregnant. Given the study's focus on interventions for reducing alcohol use during pregnancy, men and non-pregnant individuals are not eligible.
Enrollment: 40 (Estimated)
Dates: Start 2025-02-10 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Self-Reported Alcohol Consumption assessed using the Alcohol Timeline Follow Back (TLFB) | Changes from Baseline to Post Intervention in 6 weeks
  Alcohol use will be assessed using the Alcohol Timeline Follow Back (TLFB) method, a retrospective self-report tool that estimates daily drinking volume over the past month. This method provides a structured recall of alcohol consumption patterns, allowing for detailed quantification of drinking behavior.

SECONDARY OUTCOMES:
Biological Marker of Alcohol Use assessed using Phosphatidylethanol (PeTH) testing | Changes from Baseline to Post Intervention in 6 weeks
  Phosphatidylethanol (PeTH) testing, a highly specific and sensitive biomarker for alcohol consumption, will be conducted via finger-prick blood samples. PeTH levels differentiate heavy vs. occasional drinking over the past 2-3 weeks and detect recent abstinence. Dried Blood Spots (DBS) will be exported for analysis at the United States Drug Testing Laboratories (USDTL) under an established material transfer agreement, ensuring high-standard laboratory processing.
Psychosocial functioning assessed using WHO-Disability Assessment Schedule (WHO-DAS) | Changes from Baseline to Post Intervention in 6 weeks
  Measured using the WHO-Disability Assessment Schedule (WHO-DAS) evaluates functional impairment across multiple life domains, including cognition, mobility, self-care, and social participation.
Depressive Symptoms assessed using Edinburgh Postnatal Depression Scale (EPDS) | Changes from Baseline to Post Intervention in 6 weeks
  Assessed using the Edinburgh Postnatal Depression Scale (EPDS), a validated screening tool for detecting perinatal depression in pregnant women. Higher scores indicate greater symptom severity, informing potential mental health support needs.
Alcohol-Related Consequences assessed using Alcohol Use Disorder Identification Test - Consumption (AUDIT-C) | Changes from Baseline to Post Intervention in 6 weeks
  Measured using the Alcohol Use Disorder Identification Test - Consumption (AUDIT-C), a validated screening tool for identifying hazardous drinking patterns and assessing alcohol-related harm during pregnancy.

CONTACTS AND LOCATIONS:
Overall Officials: Daniela C Fuhr, Prof., Principal Investigator — Leibniz Institute for Prevention Research and Epidemiology - BIPS GmbH; Patel Peterson Williams, Prof., Principal Investigator — Medical Research Council, South Africa
Locations (1):
- South African Medical Research Council (SAMRC), Cape Town, South Africa

IPD SHARING:
Plan to Share IPD: No
The data is subject to strict confidentiality agreements as per the ethical approval obtained, and sharing it publicly could compromise participant privacy.

REFERENCES:
- [Background] Wan X, Fang M, Chen T, Wang H, Zhou Q, Wei Y, Zheng L, Zhou Y, Chen K. Corrigendum to "The mechanism of low-dose radiation-induced upregulation of immune checkpoint molecule expression in lung cancer cells" [Biochem. Biophys. Res. Commun. 608 (2022 Jun 11) 102-107, doi: 10.1016/j.bbrc.2022.03.158. Epub 2022 Apr 2.PMID: 35397421]. Biochem Biophys Res Commun. 2023 Oct 26:149132. doi: 10.1016/j.bbrc.2023.149132. Online ahead of print. No abstract available. PMID 39492324
- [Background] Petersen Williams P, Erasmus J, Myers B, Nadkarni A, Fuhr DC. Community-based counselling programme for pregnant women with alcohol problems in Cape Town, South Africa: a qualitative study of the views of pregnant women and healthcare professionals. Front Psychiatry. 2023 Jul 6;14:1203835. doi: 10.3389/fpsyt.2023.1203835. eCollection 2023. PMID 37484680